CLINICAL TRIAL: NCT04322565
Title: Colchicine to Counteract Inflammatory Response in COVID-19 Pneumonia
Brief Title: Colchicine Counteracting Inflammation in COVID-19 Pneumonia
Acronym: ColCOVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Umberto Maggiore, MD, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ColCOVID-19
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Coronavirus Infections; Pneumonia, Viral
Keywords: Colchicine; Corona Virus Infection; COVID-19
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral; COVID-19 | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): Administration of Colchicine 1mg (or 0.5 mg in CKD)/day + standard of care for COVID-19 pneumonia
  Interventions: Drug: Colchicine
- Standard of care (No Intervention): Standard of care for COVID-19 pneumonia

INTERVENTIONS:
Drug: Colchicine — Cochicine 1mg/day
  Arms: Colchicine

SUMMARY:
Cytokines and chemokines are thought to play an important role in immunity and immunopathology during virus infections [3]. Patients with severe COVID-19 have higher serum levels of pro-inflammatory cytokines (TNF-α, IL-1 and IL-6) and chemokines (IL-8) compared to individuals with mild disease or healthy controls, similar to patients with SARS or MERS . The change of laboratory parameters, including elevated serum cytokine, chemokine levels, and increased NLR in infected patients are correlated with the severity of the disease and adverse outcome, suggesting a possible role for hyper-inflammatory responses in COVID-19 pathogenesis. Importantly, previous studies showed that viroporin E, a component of SARS-associated coronavirus (SARS-CoV), forms Ca2C-permeable ion channels and activates the NLRP3 inflammasome. In addition, another viroporin 3a was found to induce NLRP3 inflammasome activation . The mechanisms are unclear.

Colchicine, an old drug used in auto-inflammatory disorders (i.e., Familiar Mediterranean Fever and Bechet disease) and in gout, counteracts the assembly of the NLRP3 inflammasome, thereby reducing the release of IL-1b and an array of other interleukins, including IL-6, that are formed in response to danger signals. Recently, colchicine has been successfully used in two cases of life-threatening post-transplant capillary leak syndrome. These patients had required mechanically ventilation for weeks and hemodialysis, before receiving colchicine, which abruptly restored normal respiratory function and diuresis over 48 hrs [4].

ELIGIBILITY:
Inclusion Criteria:

* Positive nasopharyngeal swab for COVID-19, asymptomatic or paucisymptomatic, aged ≥70 years and/or with clinical risk factors for poor outcome (clinically relevant chronic lung disease, diabetes and/or heart disease) or
* symptomatic with respiratory or systemic symptoms, however clinically stable (MEWS<3) with CT imaging showing viral pneumonia and positive or pending pharyngo-nasal swab for COVID-19: Temperature 38°C and/or intensive cough, Respiratory rate < 25 /min, oxygen saturation (pulse oximetry) >95%
* Positive swab for COVID-19
* with respiratory and/or systemic symptoms and initial mild respiratory failure e with objective signs of lung involvement; the patient is in stable conditions (MEWS < 3) Temperature>38°C and or intensive cough, Respiratory rate ≥25 /min, or oxygen saturation 94- 95% in room air

Exclusion Criteria:

* Pregnant or breast feeding
* MEWS >=3
* Hepatic failure Child-Pugh C
* Enrollment in other pharmacological studies
* Ongoing treatment with colchicine
* Ongoing treatment with antiviral drugs that include ritonavir or cobicistat
* Any medical condition or disease which in the opinion of the Investigator may place the patient at unacceptable risk for study participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | Day 28
  Time to clinical improvement: defined as time from randomization to an improvement of two points from the status at randomization on a seven-category ordinary scale
Hospital discharge | Day 28
  Live discharge from the hospital (whatever comes first)

SECONDARY OUTCOMES:
Death | Day 28
  Number of death patients
Clinical status | Day 7, Day 14
  7-category ordinal scale
Mechanical ventilhation | Day 28
  Number of patients with mechanical ventilhation
Hospitalization | Day 28
  Days of hospitalization
Time from treatment initiation to death | Day 28
  Days to death from treatment initiation
Time to Negativization COVID 19 | Day 21
  negativization of two consecutive pharyngo-nasal swab 24-72 hrs apart
Fever | Day 1,4,7,14,21,28
  Time to remission of fever in patients with T>37.5°C at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Maggiore, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- Azienda Ospedaliero Universitaria di Parma, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be avaliable from July 2020 and documentation will be shared for 10 years
Access Criteria: The sponsor recognizes the importance of communicating study data and will disclose and publish the results in a suitable form regardless of outcome. The sponsor will publish the results of this study in scientific journals

REFERENCES:
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014